CLINICAL TRIAL: NCT06041282
Title: A Multicentre Randomized Controlled Trial of Manipulation Under Anesthesia and Supervised Home Rehabilitation in the Treatment of Early Adhesive Capsulitis
Brief Title: Conservative Treatment of Early Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0750
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis
Keywords: manipulation under anesthesia; supervised home rehabilitation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manipulation under anesthesia group (Experimental): The patient underwent manipulation under anesthesia
  Interventions: Procedure: manipulation under anesthesia
- Supervised home rehabilitation group (Active Comparator): The patient underwent supervised home rehabilitation
  Interventions: Procedure: supervised home rehabilitation

INTERVENTIONS:
Procedure: manipulation under anesthesia — After the anesthesia took effect, the patient was placed in the supine position, and the experienced surgeon stood at the head of the bed to release the affected limb by four angles of forward flexion, abduction, external rotation and internal rotation. After the operation is completed, 1ml de Bosson (MSD) +2.5ml sodium hyaluronate (Biochemical Industries Co., LTD.) is injected once.
  Arms: manipulation under anesthesia group
Procedure: supervised home rehabilitation — The doctor instructs the patient in exercise training at the outpatient clinic. At each clinic visit, the doctor will guide the different stages of the movement. At the first visit, the doctor guides the patient through the first phase of the rehabilitation program to improve the patient's basic mobility. At the first month of follow-up, the second phase of rehabilitation program was guided, and the recovery of mobility was accompanied by muscle training, including wall climbing and muscle resistance exercises. 1ml Debossone (MSD) +2.5ml sodium hyaluronate (Biochemical Industries Co., LTD.) was injected once at the clinic. All the training required patients to do their best at home to complete 3 sets of 5 each. At the end of each day, the patient will upload a video to the platform, and the doctor will evaluate whether the patient's recovery is in place.
  Arms: Supervised home rehabilitation group

SUMMARY:
A prospective, multicentre, randomized controlled study comparing the efficacy of conservative treatment for early adhesive capsulitis

DETAILED DESCRIPTION:
This clinical trial evaluated the most common protocols for the treatment of adhesive capsulitis in secondary hospitals. To compare the efficacy of manipulation under anesthesia and supervised home conservative treatment of early adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients in our hospital who need manual release of periarthritis of shoulder or home rehabilitation treatment;
* Unilateral and primary periarthritis of shoulder
* Age ≥40 years old and ≤80 years old, regardless of gender.
* Forward flexion movement is more than 50% limited compared with the contralateral.
* Duration of disease ≤3 months

Exclusion Criteria:

* Patients with a previous history of shoulder joint surgery
* Patients who did not complete the follow-up within the specified time
* Patients with other shoulder diseases.
* Patient with systemic immune disease.
* Patients who have participated in clinical trials or are conducting other clinical trials within 3 months before screening
* Patients with serious primary cardiovascular diseases, lung diseases, endocrine and metabolic diseases, or serious diseases affecting their survival, such as tumor or AIDS, are considered not suitable for admission.
* Patients with serious liver diseases, kidney diseases, hematological diseases, such as kidney function (BUN, Cr) more than the upper limit of normal, liver function (ALT, AST, TBIL) more than 2 times the upper limit of normal.
* Patients with viral hepatitis, infectious diseases, abnormal blood coagulation mechanism and other diseases that researchers consider inappropriate for surgery.
* Pregnant or lactating women, or those planning to get pregnant during the test, with positive urine HCG test results before the test; Menstruating women should wait until their period is over before undergoing surgery.
* Patients with severe neurological and mental diseases.
* Suspected or true history of alcohol and drug abuse.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score (CMS) | 6months after intervention
  The Constant-Mulery score mainly includes 8 aspects related to your shoulder in the past 4 weeks.
  The proportion of subjective and objective components in the Constant-Mulery score is 35 points/65 points. A total of 100 points.The subjective part of the score includes the score of pain degree and the score of impact on daily life. 35 points in total.The objective part of the score includes the score of shoulder range of motion and strength. 65 points in total.

SECONDARY OUTCOMES:
Constant-Murley Score (CMS) | 1 months, 3months, and 1year after intervention
  The Constant-Mulery score mainly includes 8 aspects related to your shoulder in the past 4 weeks.
  The proportion of subjective and objective components in the Constant-Mulery score is 35 points/65 points. A total of 100 points.The subjective part of the score includes the score of pain degree and the score of impact on daily life. 35 points in total.The objective part of the score includes the score of shoulder range of motion and strength. 65 points in total.
Oxford Shoulder Score (OSS) | 1 months, 3months, 6 months and 1year after intervention
  The Oxford Shoulder Score (OSS) consists of 12 questions with five options each. The light to heavy lines were assigned 1, 2, 3, 4 and 5 points respectively. So the total score is between 12 and 60. A score of 12 represents perfectly normal shoulder function and a score of 60 represents the most severe difficulty in shoulder function.
Fear-avoidance belief questionnaire(FABQ) | 1 months, 3months, 6 months and 1year after intervention
  The FABQ is a self-assessment scale with 16 options. Each option has 0~6 points and 7 grades (from extremely disagreeable to extremely agreed). "0" means completely disagreed, "6" means completely agreed, and "1~5" means not sure. The higher the score, the more inclined to fully agree
Insomnia Severity Index(ISI) | 1 months, 3months, 6 months and 1year after intervention
  The scale is a simple tool for screening insomnia, including 7 items, which are used to evaluate the nature and symptoms of sleep disorders of subjects.
Hospital Anxiety and Depression Scale(HADS) | 1 months, 3months, 6 months and 1year after intervention
  HADS is a self-assessment scale, including two subscales, HADS-A and HADS-D, with a total of 14 items, including 7 items for anxiety (A) and 7 items for depression (D). Each item is scored at four levels according to the frequency of symptoms in the past month. Each item is scored at 0-3 points in four levels. The higher the score, the more serious the anxiety or depression
SF-36 | 1 months, 3months, 6 months and 1year after intervention
  SF-36 is a concise health questionnaire developed by the Boston Institute of Health, which is widely used in the measurement of the quality of life of the general population, the evaluation of clinical trials and the evaluation of health policies. SF-36 is used to assess physiological function, physiological function, physical pain, general health, energy, social function, emotional function and mental health, which are classified into "physical health" and "mental health"
Visual analogue scale(VAS) | 1 months, 3months, 6 months and 1year after intervention
  Draw a 10cm horizontal line on the paper. One end of the line is "0", indicating no pain; the other end is "10", indicating severe pain; The middle represents different degrees of pain; Let the patient draw a mark on the horizontal line according to their feelings to indicate the degree of pain.
range of motion | 1 months, 3months, 6 months and 1year after intervention
  Measure the patient's flexion, abduction, internal rotation and external rotation angle

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China